CLINICAL TRIAL: NCT04942379
Title: Asthma Link: A Real World Application of School Supervised Asthma Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michelle Trivedi, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H00016378; 5K23HL150341 (NIH)
Record Dates: First submitted 2021-05-12; First posted 2021-06-28 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Childhood Asthma
Keywords: asthma; childhood asthma; stakeholder engagement; medication adherence; school-supervised asthma therapy; real-world; pragmatic trial
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma Link (Experimental): Site providers will be trained to efficiently discuss school-supervised medication administration with families and school nurses. Providers identify children with poorly controlled asthma and poor medication adherence and offer enrollment in Asthma Link to provide school-supervised asthma therapy. Ongoing communication occurs between the pediatric practice, school nurse and families through electronic medical record messaging and phone communication. Data will be collected at baseline (study entry) and at 3-, 6-and 12-month follow-up.
  Interventions: Other: Asthma Link
- Enhanced Usual Care (Active Comparator): Sites will receive pediatric pulmonologist-delivered training and a workbook for pediatric practices to provide to patients on behavioral strategies to help promote asthma medication adherence. Providers identify children with poorly controlled asthma and poor medication adherence and offer enrollment to this Enhanced Usual Care condition of study (receipt of workbook). Data will also be collected at baseline (study entry) and at 3-, 6-and 12-month follow-up.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: Asthma Link — Providers enroll patients in school nurse supervised daily controller asthma medication delivery
  Arms: Asthma Link
Other: Enhanced Usual Care — Providers counsel patients on behavioral strategies to improve medication adherence. Patients also receive an asthma workbook outlining behavioral strategies for asthma medication adherence.
  Arms: Enhanced Usual Care

SUMMARY:
The goal of this study is to assess the feasibility of a clinical trial to evaluate the impact and process of deploying school-supervised asthma therapy in a real-world setting for children with poorly controlled asthma (aged 6-17 years).

DETAILED DESCRIPTION:
The proposed 4-site pilot cluster randomized controlled trial will assess the feasibility of conducting a clinical trial of Asthma Link, a real-world school-supervised asthma therapy program. We will compare the impact of Asthma Link deployed in 2 pediatric practice sites versus Enhanced usual care deployed in 2 comparator sites, with 18 parent-child dyads enrolled per site (N=72 dyads).

Primary trial outcomes will be participant recruitment, retention, and intervention fidelity. Secondary trial outcomes will be differences in the frequency of asthma symptoms, emergency department visits, hospital admissions, courses of oral corticosteroids, spirometry values, medication adherence and school absences between intervention and enhanced usual care sites at 3, 6 and 12 month follow up. Additionally we will assess process outcomes (acceptability, adoption, costs, sustainability).

ELIGIBILITY:
STUDY INCLUSION/EXCLUSION CRITERIA:

Child Inclusion Criteria:

* Meet the eligibility criteria for Asthma Link (as described below)
* Enrolled in Asthma Link (if randomized to the Asthma Link Condition)
* Able and willing to provide informed assent

Child Exclusion Criteria:

* Unable or unwilling to provide informed assent
* Diagnosis of a serious co-morbid illness during the past 5 years
* Developmental delay that would prevent study participation.
* Planning on moving from primary residence or moving outside of the school district in the next 1 year
* A sibling to a child participating in this study

Parent Inclusion Criteria:

* Parent/guardian to patient
* 18 years or older
* Able to understand and communicate in English or Spanish
* Able and willing to provide informed consent.

Parent Exclusion Criteria:

* Adults lacking capacity
* Prisoners

Medical Provider, School Nurse, Asthma Champion Inclusion Criteria:

• Able and willing to provide informed consent

Medical Provider, School Nurse, Asthma Champion Exclusion Criteria:

• Unable or unwilling to provide informed consent

Child eligibility for children enrolled in Asthma Link:

* children aged 6-17 years (enrolled in grade 1-12)
* prescribed daily inhaled corticosteroid (ICS) for asthma
* 1 or more courses of oral steroids in the past 2 years OR 1 or more hospitalizations or ED visits for asthma in the past 2 years OR 1 or more sick visits for asthma in the past year OR Asthma Control Test (ACT) score <19
* parent/child report of poor ICS adherence on adherence checklist- i.e. child or parent says "Yes" when provider asks if they have difficulty remembering to take their medication or if they regularly take medication holidays or breaks
* able and willing to assent
* parental permission
* English or Spanish speaking

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Trivedi, MD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- University of Massachusetts, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asthma Link | Enhanced Usual Care
Started | 31 | 35
3 Months | 29 | 34
6 Months | 28 | 32
Completed (12 months) | 27 | 32
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asthma Link | Enhanced Usual Care | Total
Number analyzed (Participants) | 31 | 35 | 66
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 31 | 35 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 17 | 15 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 20 | 43
  Not Hispanic or Latino | 8 | 15 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 8 | 15 | 23
  More than one race | 8 | 5 | 13
  Unknown or Not Reported | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Procedures Assessed by Number of Patients Screened
Description: Research staff will track number of patients screened during enrollment process.
Time Frame: Baseline
Population: These numbers reflect the total number of patients screened for eligibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Link | Enhanced Usual Care
Number analyzed (Participants) | 143 | 208
Participants | 143 | 208

2. Primary Outcome: Recruitment Procedures Assessed by Number of Eligible Participants
Description: Research staff will track number of eligible participants who meeting study criteria during the enrollment process.
Time Frame: Baseline
Population: These numbers reflect the number of participants who were eligible based on initial screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Link | Enhanced Usual Care
Number analyzed (Participants) | 143 | 208
Participants | 66 | 55

3. Primary Outcome: Recruitment Procedures Assessed by Number of Patients Recruited Into the Study
Description: Research staff will track number of patients recruited into the study after they are assessed for eligibility.
Time Frame: Baseline
Population: Overall number of participants analyzed reflects the number of participants who were eligible on initial screen.
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Link | Enhanced Usual Care
Number analyzed (Participants) | 66 | 55
Participants | 31 | 35

4. Primary Outcome: Recruitment Procedures Assessed by Number of Eligible Patients That Were Not Enrolled or Refused to Participate.
Description: Research staff will track the number of patients that were not enrolled or refused to participate in the study along with the reasons for non-enrollment.
Time Frame: Baseline
Population: These numbers reflect the number of eligible participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Link | Enhanced Usual Care
Number analyzed (Participants) | 66 | 55
Participants | 35 | 20

5. Primary Outcome: Retention of Study Participants (Drop Out)
Description: Research staff to track number of participants who drop out of the study and note reasons for not completing study.
Time Frame: Up to end of study, approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Link | Enhanced Usual Care
Number analyzed (Participants) | 31 | 35
Participants | 0 | 0

6. Primary Outcome: Retention of Study Participants (Lost to Follow-up)
Description: Research staff to track number of participants lost to follow-up, who did not complete the 12 month study assessment.
Time Frame: Up to end of study, approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Link | Enhanced Usual Care
Number analyzed (Participants) | 31 | 35
Participants | 4 | 3

7. Primary Outcome: Intervention Fidelity - Pediatric Practice
Description: Research staff to assess for intervention fidelity within the pediatric practice through a checklist for pediatric staff to assess percentage of eligible children enrolled.
Time Frame: Baseline
Population: These numbers reflect the number of patients eligible for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Link | Enhanced Usual Care
Number analyzed (Participants) | 66 | 55
Participants | 31 | 35

8. Primary Outcome: Intervention Fidelity - Percentage of Enrolled Students Receiving Intervention
Description: Research staff to assess for intervention fidelity by school nurse report of percentage of enrolled students receiving supervised therapy.
Time Frame: Up to end of study, approximately 12 months
Population: Participants in the Enhanced Usual Care group did not receive school supervised therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Link | Enhanced Usual Care
Number analyzed (Participants) | 31 | 0
Participants | 31 | 0

9. Primary Outcome: Intervention Fidelity - School Nurse and Family Participation
Description: Research staff to assess for intervention fidelity by school nurse checklist of each enrolled child attending daily school nurse sessions and his/her family bringing medication to school.
Time Frame: Up to end of study, approximately 12 months
Population: Participants in the Enhanced Usual Care group did not receive school supervised therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma Link | Enhanced Usual Care
Number analyzed (Participants) | 31 | 0
Participants | 31 | 0

10. Secondary Outcome: Acceptability - Participants
Description: Research staff will assess acceptability of the study among stakeholders (parent-child dyads, medical providers, school nurses) via a survey in which we will ask stakeholders to rate each component of the Asthma Link intervention using a study specific Acceptability scale ranging from 1 (strongly disagree) to 5 (strongly agree). Qualitative interviews will be performed with stakeholders at 12 months
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

11. Secondary Outcome: Adoption of Asthma Link Intervention - Medical Provider
Description: Research staff will assess adoption of the intervention via Pediatric practice log to track number of providers offering Asthma Link.
Time Frame: Baseline, 3 months, 6 months, 12 months
Reporting Status: Not Posted

12. Secondary Outcome: Adoption of Asthma Link Intervention - Participant
Description: Research staff will assess adoption of the intervention via survey to family at each survey timepoint of study to assess ability to obtain 2 inhalers (one for home and one for school) and deliver medicine to school.
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

13. Secondary Outcome: Adoption of Asthma Link Intervention - School Nurse
Description: Research staff will assess adoption of the intervention via school nurse log to track family bringing in medicine to school and frequency of child coming to nurses office to receive the medication.
Time Frame: Baseline, 3 months, 6 months, 12 months
Reporting Status: Not Posted

14. Secondary Outcome: Cost Effectiveness of Intervention
Description: Research staff will use survey questions to assess time and costs for school nurses to review the toolkit and administer the intervention, pediatric providers to implement the program, and parents to participate in the intervention
Time Frame: School nurses and pediatric practices 6 and 12 months/Parents 3, 6 and 12 months
Reporting Status: Not Posted

15. Secondary Outcome: Sustainability of Intervention
Description: Research staff will use a survey questions to parents, pediatric practice staff and school staff
Time Frame: 3 months, 6 months, 12 months
Reporting Status: Not Posted

16. Secondary Outcome: Asthma Symptoms - Spirometry
Description: Research staff will assess asthma symptoms utilizing spirometry to measure Forced Expiratory Volume.
Time Frame: Baseline, 3 months, 6 months, 12 months
Reporting Status: Not Posted

17. Secondary Outcome: Asthma Symptoms - Asthma Control Test
Description: Research staff will assess asthma symptoms utilizing the validated measure: Asthma Control Test (ACT) which consists of parent's assessment of level of control over child's asthma symptoms in the previous 4 weeks.
Time Frame: Baseline, 3 months, 6 months, 12 months
Reporting Status: Not Posted

18. Secondary Outcome: Asthma Symptoms - Maximum Symptoms Days
Description: Research staff will assess asthma symptoms utilizing the validated measure: Maximum Symptom Days (the largest value of the number of days in the previous 2 weeks that a parent reports that their child experienced a) cough, wheezing, or shortness of breath, b) slowed activities due to symptoms, or 3)nocturnal awakening due to these symptoms.
Time Frame: Baseline, 3 months, 6 months, 12 months
Reporting Status: Not Posted

19. Secondary Outcome: Frequency of Healthcare Utilization Over Time
Description: Research staff will assess the frequency of healthcare utilization (# of emergency room visits, # of hospital admissions, # of oral steroid courses, and # of urgent care visits) due to asthma through parent report on surveys and medical record review.
Time Frame: Baseline, 3 months, 6 months, 12 months
Reporting Status: Not Posted

20. Secondary Outcome: Medication Adherence
Description: Research staff will assess medication adherence via a survey questions administered to parents and through pharmacy refill data.
Time Frame: Baseline, 3 months, 6 months, 12 months
Reporting Status: Not Posted

21. Secondary Outcome: School Absences
Description: Research staff will assess school absences via parent report and school nurse report
Time Frame: Baseline, 3 months, 6 months, 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of the 12 months participants were in the study.
Arm/Group | Asthma Link | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/35
Other Adverse Events (participants affected / at risk) | 0/31 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT04942379/Prot_SAP_000.pdf